CLINICAL TRIAL: NCT05002283
Title: Accuracy of Computer Guided Free Gingival Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Shawky, Principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS 3-3-5
Record Dates: First submitted 2021-08-01; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Computer Guided; Free Gingival Graft

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): the patients undergo free gingival graft harvest from the palate using a patient specific guide
  Interventions: Other: patient specific guide

INTERVENTIONS:
Other: patient specific guide — harvesting palatal free gingival graft using the patient specific guide

SUMMARY:
A patient specific surgical guide for harvesting of free gingival graft from the palate

ELIGIBILITY:
Inclusion Criteria:

* patients with intraoral alveolar defect requiring soft tissue augmentation

Exclusion Criteria:

1. - patients with systemic diseases interfering with surgical interventions
2. - Poor oral hygiene

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of the guide | One month
  accuracy of the predefined graft dimensions relative to the required dimensions of the recipient site in millimetres

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shawky, MSc, Principal Investigator — Investigator
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
the IPD will be made available upon request from the author